CLINICAL TRIAL: NCT00125593
Title: Study of Heart and Renal Protection (SHARP): The Effects of Lowering LDL-cholesterol With Simvastatin 20mg Plus Ezetimibe 10mg in Patients With Chronic Kidney Disease: a Randomized Placebo-controlled Trial
Brief Title: Study of Heart and Renal Protection
Acronym: SHARP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Schering-Plough (Industry); National Health and Medical Research Council, Australia (Other); British Heart Foundation (Other); Medical Research Council (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CTSUSHARP1; ISRCTN54137607 (Other: ISRCTN (Current Controlled Trials)); EudraCT - 2004-001156-37 (Other: European Union); UK CRN 2542 (Other: United Kingdom Clinical Research Network)
Record Dates: First submitted 2005-07-29; First posted 2005-08-01 (Estimated); Results first posted 2012-02-01 (Estimated); Last update posted 2012-02-01 (Estimated); Status verified 2012-01

CONDITIONS: Kidney Disease, Chronic
Keywords: Kidney Disease, Chronic; LDL cholesterol; simvastatin; ezetimibe; cardiovascular disease; atherosclerosis
MeSH Terms: conditions — Renal Insufficiency, Chronic; Cardiovascular Diseases; Atherosclerosis | interventions — Simvastatin; Ezetimibe; Ezetimibe, Simvastatin Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Placebo = Arm 1. A double-dummy method ensured that patients and study staff were unaware of the treatment allocation, with all Arm 1 patients taking 2 tablets (placebo simvastatin plus ezetimibe tablet with a placebo simvastatin tablet) during the first year. After the first year, all Arm 1 patients took one tablet (placebo simvastatin plus ezetimibe tablet).
  Interventions: Drug: Placebo
- Simvastatin 20mg plus Ezetimibe 10mg (Active Comparator): Simvastatin 20mg plus ezetimibe 10mg = Arm 2. A double-dummy method ensured that patients and study staff were unaware of the treatment allocation, with all Arm 2 patients taking 2 tablets during the first year (active simvastatin plus ezetimibe tablet with a placebo simvastatin tablet). After the first year, all Arm 2 patients took one tablet (active simvastatin 20mg plus ezetimibe 10mg tablet).
  Interventions: Drug: Simvastatin 20 mg; Drug: Ezetimibe 10mg
- Simvastatin 20mg (Other): Simvastatin 20mg alone = Arm 3. After 1 year, those initially allocated to Arm 3 were re-randomized to simvastatin 20mg plus ezetimibe 10mg (Arm 3b) daily or placebo (Arm 3a). A double-dummy method ensured that patients and study staff were unaware of the treatment allocation, with Arm 3 patients taking 2 tablets (a placebo simvastatin plus ezetimibe tablet with an active simvastatin tablet) during the first year. After the first year, all Arm 3a and Arm 3b patients took one tablet (active or placebo simvastatin plus ezetimibe tablet).
  Interventions: Drug: Simvastatin 20 mg

INTERVENTIONS:
Drug: Simvastatin 20 mg — Once daily
  Other Names: Zocor
  Arms: Simvastatin 20mg; Simvastatin 20mg plus Ezetimibe 10mg
Drug: Ezetimibe 10mg — Once daily
  Other Names: Ezetrol; Zetia; Vytorin (simvastatin plus ezetimibe)
  Arms: Simvastatin 20mg plus Ezetimibe 10mg
Drug: Placebo — Once daily
  Arms: Placebo

SUMMARY:
The chief aim of SHARP was to determine whether lowering blood LDL cholesterol with simvastatin (20mg) plus ezetimibe (10mg) daily could safely reduce the risk of coronary heart disease, non-hemorrhagic stroke and the need for revascularization procedures in patients with chronic kidney disease (CKD). It also aimed to assess whether lowering LDL cholesterol reduced the rate of loss of renal function in people with CKD who had not commenced dialysis treatment.

DETAILED DESCRIPTION:
The SHARP (Study of Heart and Renal Protection) was a double-blind placebo-controlled trial which aimed to assess the safety and efficacy of reducing LDL cholesterol in more than 9,000 patients with chronic kidney disease (about 3,000 of whom were on dialysis at randomization).

Patients were randomly assigned to simvastatin 20 mg plus ezetimibe 10 mg daily versus matching placebo (a subset of these patients had previously received simvastatin 20mg only and were then randomly re-assigned to receive simvastatin 20mg plus ezetimibe 10mg or placebo at one year). Details of the SHARP trial design and methods have been reported previously (reference: Am Heart J 2010; 160:785-94.).

SHARP was overseen by an independent Steering Committee that included nephrologists, cardiologists, clinical trialists, and statisticians, with 2 non-voting observers from the main funder (Merck/Schering-Plough Pharmaceuticals). The independent sponsor was the University of Oxford, and the trial was funded by Merck/Schering-Plough Pharmaceuticals, the Australian National Health and Medical Research Council, the British Heart Foundation and the UK Medical Research Council.

In October 2009, the Steering Committee decided (blind to the effects of study treatment on clinical outcomes) to change the original protocol-specified primary outcome to a revised key outcome of major atherosclerotic events, defined as the combination of non-fatal myocardial infarction, coronary death, ischemic stroke, or any revascularization procedure (i.e. exclusion of non-coronary cardiac deaths and strokes confirmed to be hemorrhagic from the original major vascular event outcome). These and other changes are described in the revised statistical analysis plan for SHARP (reference: Am Heart J 2010; 160:785-94.). Accordingly, the chief emphasis of the published results (reference: Lancet 2011; 377:2181-92) is on the revised pre-specified key outcome of first major atherosclerotic events.

ELIGIBILITY:
Inclusion Criteria:

* History of chronic kidney disease (CKD): either patients who are pre-dialysis (with a plasma or serum creatinine greater than or equal to 150 micromol/l [greater than or equal to 1.7 mg/dl] in men, or greater than or equal to 130 micromol/l [greater than or equal to 1.5 mg/dl] in women); or patients on dialysis (hemodialysis or peritoneal dialysis)
* Men or women aged greater than or equal to 40 years

Exclusion Criteria:

* Definite history of myocardial infarction or coronary revascularization procedure
* Functioning renal transplant, or living donor-related transplant planned
* Less than 2 months since presentation as an acute uraemic emergency (but could be entered later, if appropriate)
* Definite history of chronic liver disease, or abnormal liver function (i.e. alanine aminotransferase [ALT] greater than 1.5 x upper limit of normal [ULN] or, if ALT not available, aspartate aminotransferase [AST] greater than 1.5 x ULN). (Note: Patients with a history of hepatitis were eligible provided these limits were not exceeded.)
* Evidence of active inflammatory muscle disease (e.g. dermatomyositis, polymyositis), or creatine kinase (CK) greater than 3 x ULN
* Definite previous adverse reaction to a statin or to ezetimibe
* Concurrent treatment with a contraindicated drug. (Note: Patients who were temporarily taking such drugs could have been re-screened for participation in the study when they discontinued them, if appropriate.) These contraindicated drugs included: HMG-CoA reductase inhibitor ("statin"); fibric acid derivative ("fibrate"); nicotinic acid; macrolide antibiotic (erythromycin, clarithromycin); systemic use of imidazole or triazole antifungals (e.g. itraconazole, ketoconazole); protease-inhibitors (e.g. antiretroviral drugs for HIV infection); nefazodone; ciclosporin
* Child-bearing potential (i.e. premenopausal woman who was not using a reliable method of contraception)
* Known to be poorly compliant with clinic visits or prescribed medication
* Medical history that might have limited the individual's ability to take trial treatments for the duration of the study (e.g. severe respiratory disease, history of cancer other than non-melanoma skin cancer, or recent history of alcohol or substance misuse)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9438 (Actual)
Dates: Start 2003-06; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Colin Baigent, FRCP, FFPH, Principal Investigator — Clinical Trial Service Unit & Epidemiological Studies Unit, University of Oxford; Martin J Landray, PhD, FRCP, Principal Investigator — Clinical Trial Service Unit & Epidemiological Studies Unit, University of Oxford
Locations (1):
- Clinical Trial Service Unit & Epidemiological Studies Unit, University of Oxford, Oxford, United Kingdom

REFERENCES:
- [Background] Baigent C, Landray M, Leaper C, Altmann P, Armitage J, Baxter A, Cairns HS, Collins R, Foley RN, Frighi V, Kourellias K, Ratcliffe PJ, Rogerson M, Scoble JE, Tomson CR, Warwick G, Wheeler DC. First United Kingdom Heart and Renal Protection (UK-HARP-I) study: biochemical efficacy and safety of simvastatin and safety of low-dose aspirin in chronic kidney disease. Am J Kidney Dis. 2005 Mar;45(3):473-84. doi: 10.1053/j.ajkd.2004.11.015. PMID 15754269
- [Background] Landray M, Baigent C, Leaper C, Adu D, Altmann P, Armitage J, Ball S, Baxter A, Blackwell L, Cairns HS, Carr S, Collins R, Kourellias K, Rogerson M, Scoble JE, Tomson CR, Warwick G, Wheeler DC. The second United Kingdom Heart and Renal Protection (UK-HARP-II) Study: a randomized controlled study of the biochemical safety and efficacy of adding ezetimibe to simvastatin as initial therapy among patients with CKD. Am J Kidney Dis. 2006 Mar;47(3):385-95. doi: 10.1053/j.ajkd.2005.11.018. PMID 16490616
- [Background] Sharp Collaborative Group. Study of Heart and Renal Protection (SHARP): randomized trial to assess the effects of lowering low-density lipoprotein cholesterol among 9,438 patients with chronic kidney disease. Am Heart J. 2010 Nov;160(5):785-794.e10. doi: 10.1016/j.ahj.2010.08.012. Epub 2010 Sep 18. PMID 21095263
- [Result] Baigent C, Landray MJ, Reith C, Emberson J, Wheeler DC, Tomson C, Wanner C, Krane V, Cass A, Craig J, Neal B, Jiang L, Hooi LS, Levin A, Agodoa L, Gaziano M, Kasiske B, Walker R, Massy ZA, Feldt-Rasmussen B, Krairittichai U, Ophascharoensuk V, Fellstrom B, Holdaas H, Tesar V, Wiecek A, Grobbee D, de Zeeuw D, Gronhagen-Riska C, Dasgupta T, Lewis D, Herrington W, Mafham M, Majoni W, Wallendszus K, Grimm R, Pedersen T, Tobert J, Armitage J, Baxter A, Bray C, Chen Y, Chen Z, Hill M, Knott C, Parish S, Simpson D, Sleight P, Young A, Collins R; SHARP Investigators. The effects of lowering LDL cholesterol with simvastatin plus ezetimibe in patients with chronic kidney disease (Study of Heart and Renal Protection): a randomised placebo-controlled trial. Lancet. 2011 Jun 25;377(9784):2181-92. doi: 10.1016/S0140-6736(11)60739-3. Epub 2011 Jun 12. PMID 21663949
- [Derived] Tunnicliffe DJ, Palmer SC, Cashmore BA, Saglimbene VM, Krishnasamy R, Lambert K, Johnson DW, Craig JC, Strippoli GF. HMG CoA reductase inhibitors (statins) for people with chronic kidney disease not requiring dialysis. Cochrane Database Syst Rev. 2023 Nov 29;11(11):CD007784. doi: 10.1002/14651858.CD007784.pub3. PMID 38018702
- [Derived] Sukkar L, Talbot B, Jun M, Dempsey E, Walker R, Hooi L, Cass A, Jardine M, Gallagher M. Protocol for the Study of Heart and Renal Protection-Extended Review: Additional 5-Year Follow-up of the Australian, New Zealand, and Malaysian SHARP Cohort. Can J Kidney Health Dis. 2019 Oct 14;6:2054358119879896. doi: 10.1177/2054358119879896. eCollection 2019. PMID 31662874
- [Derived] Schlackow I, Kent S, Herrington W, Emberson J, Haynes R, Reith C, Collins R, Landray MJ, Gray A, Baigent C, Mihaylova B; SHARP Collaborative Group. Cost-effectiveness of lipid lowering with statins and ezetimibe in chronic kidney disease. Kidney Int. 2019 Jul;96(1):170-179. doi: 10.1016/j.kint.2019.01.028. Epub 2019 Mar 12. PMID 31005271
- [Derived] Schlackow I, Kent S, Herrington W, Emberson J, Haynes R, Reith C, Wanner C, Fellstrom B, Gray A, Landray MJ, Baigent C, Mihaylova B; SHARP Collaborative Group. A policy model of cardiovascular disease in moderate-to-advanced chronic kidney disease. Heart. 2017 Dec;103(23):1880-1890. doi: 10.1136/heartjnl-2016-310970. Epub 2017 Aug 5. PMID 28780579
- [Derived] Reith C, Staplin N, Herrington WG, Stevens W, Emberson J, Haynes R, Mafham M, Armitage J, Cass A, Craig JC, Jiang L, Pedersen T, Baigent C, Landray MJ; SHARP Collaborative Group. Effect on non-vascular outcomes of lowering LDL cholesterol in patients with chronic kidney disease: results from the Study of Heart and Renal Protection. BMC Nephrol. 2017 May 1;18(1):147. doi: 10.1186/s12882-017-0545-2. PMID 28460629
- [Derived] Herrington W, Staplin N, Judge PK, Mafham M, Emberson J, Haynes R, Wheeler DC, Walker R, Tomson C, Agodoa L, Wiecek A, Lewington S, Reith CA, Landray MJ, Baigent C; SHARP Collaborative Group. Evidence for Reverse Causality in the Association Between Blood Pressure and Cardiovascular Risk in Patients With Chronic Kidney Disease. Hypertension. 2017 Feb;69(2):314-322. doi: 10.1161/HYPERTENSIONAHA.116.08386. Epub 2016 Dec 27. PMID 28028192
- [Derived] Morton RL, Schlackow I, Staplin N, Gray A, Cass A, Haynes R, Emberson J, Herrington W, Landray MJ, Baigent C, Mihaylova B; SHARP Collaborative Group. Impact of Educational Attainment on Health Outcomes in Moderate to Severe CKD. Am J Kidney Dis. 2016 Jan;67(1):31-9. doi: 10.1053/j.ajkd.2015.07.021. Epub 2015 Sep 16. PMID 26385817
- [Derived] Peto R, Emberson J, Landray M, Baigent C, Collins R, Clare R, Califf R. Analyses of cancer data from three ezetimibe trials. N Engl J Med. 2008 Sep 25;359(13):1357-66. doi: 10.1056/NEJMsa0806603. Epub 2008 Sep 2. PMID 18765432
- See also: SHARP homepage — http://www.ctsu.ox.ac.uk/~sharp/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: SHARP was conducted in 380 centres in 18 countries: Austria, Australia, Canada, China, The Czech Republic, Denmark, Finland, France, Germany, Malaysia, The Netherlands, New Zealand, Norway, Poland, Sweden, Thailand, the United Kingdom and the United States of America. Recruitment occurred between 2003 and 2006.
Pre-assignment Details: Run-in period between screening and randomization of ~ 6 weeks duration. 11792 patients screened and 9438 randomized to the initial 3 arms. Overall 9270 patients were randomly assigned to simvastatin plus ezetimibe (4650 patients, 4193 initially plus 457 after first year) versus placebo (4620 patients, 4191 initially plus 429 after first year).
Groups:
- Simvastatin 20mg Plus Ezetimibe 10mg: A double-dummy method ensured that patients and study staff were unaware of the treatment allocation, with all patients taking 2 tablets during the first year (active simvastatin plus ezetimibe tablet with a placebo simvastatin tablet). After the first year, all patients took one tablet (active simvastatin 20mg plus ezetimibe 10mg tablet).
- Placebo: A double-dummy method ensured that patients and study staff were unaware of the treatment allocation, with all patients taking 2 tablets (placebo simvastatin plus ezetimibe tablet with a placebo simvastatin tablet) during the first year. After the first year, all patients took one tablet (placebo simvastatin plus ezetimibe tablet).
Period: Overall Study
Arm/Group | Simvastatin 20mg Plus Ezetimibe 10mg | Placebo
Started | 4650 | 4620
Completed | 4549 | 4517
Not Completed | 101 | 103

BASELINE CHARACTERISTICS:
Groups:
- Simvastatin Plus Ezetimibe; Placebo: Once daily tablet
- Total: Total of all reporting groups
Arm/Group | Simvastatin Plus Ezetimibe | Placebo | Total
Number analyzed (Participants) | 4650 | 4620 | 9270
Age Continuous [Mean (Standard Deviation); unit: Years] | 62 (12) | 62 (12) | 62 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1735 | 1735 | 3470
  Male | 2915 | 2885 | 5800
Renal status [Number; unit: Participants]
  On dialysis | 1533 | 1490 | 3023
  Not on dialysis | 3117 | 3130 | 6247

OUTCOME MEASURES:

1. Primary Outcome: Key Outcome as Per Statistical Analysis Plan = Major Atherosclerotic Events Among All Patients Ever Randomized to Simvastatin Plus Ezetimibe Versus All Patients Allocated to Placebo
Description: Major atherosclerotic events defined as non-fatal myocardial infarction or coronary death, non-hemorrhagic stroke, or any arterial revascularization procedure (excluding dialysis access procedures). Numbers provided = number of patients with events.
Time Frame: Median follow-up 4.9 years
Measure: Number; unit: participants
Groups:
- Simvastatin Plus Ezetimibe: A double-dummy method ensured that patients and study staff were unaware of the treatment allocation, with all patients taking 2 tablets during the first year (active simvastatin plus ezetimibe tablet with a placebo simvastatin tablet). After the first year, all patients took one tablet (active simvastatin 20mg plus ezetimibe 10mg tablet).
Arm/Group | Simvastatin Plus Ezetimibe | Placebo
Number analyzed (Participants) | 4650 | 4620
participants | 526 | 619
Statistical Analysis 1: Comparison: Simvastatin Plus Ezetimibe vs Placebo; All analyses by intention to treat; Test type: Superiority or Other; p = 0.0021, Log Rank; Risk Ratio (RR) = 0.83, 95% CI 2-sided [0.74 to 0.94]

2. Secondary Outcome: Major Vascular Events Analyzed Among All Patients Ever Randomized to Simvastatin Plus Ezetimibe Versus All Patients Allocated to Placebo
Description: Major vascular events defined as non-fatal myocardial infarction or cardiac death, any stroke, or any arterial revascularization procedure (excluding dialysis access procedures). Numbers provided = number of patients with events.
Time Frame: Median follow-up 4.9 years
Measure: Number; unit: participants
Arm/Group | Simvastatin Plus Ezetimibe | Placebo
Number analyzed (Participants) | 4650 | 4620
participants | 701 | 814
Statistical Analysis 1: Comparison: Simvastatin Plus Ezetimibe vs Placebo; All analyses by intention to treat; Test type: Superiority or Other; p = 0.0012, Log Rank; Risk Ratio (RR) = 0.85, 95% CI 2-sided [0.77 to 0.94]

3. Secondary Outcome: Major Vascular Events Analyzed Amongst Patients Initially Randomized to Simvastatin Plus Ezetimibe Versus Placebo (Original Protocol-defined Primary Outcome)
Description: as for outcome 2
Time Frame: Median follow-up 4.9 years
Population: Includes only those patients initially randomized to simvastatin plus ezetimibe versus placebo (as opposed to all patients ever randomized to simvastatin plus ezetimibe versus all patients allocated placebo)
Measure: Number; unit: participants
Arm/Group | Simvastatin Plus Ezetimibe | Placebo
Number analyzed (Participants) | 4193 | 4191
participants | 639 | 749
Statistical Analysis 1: Comparison: Simvastatin Plus Ezetimibe vs Placebo; All analyses by intention to treat; Test type: Superiority or Other; p = 0.001, Log Rank; Risk Ratio (RR) = 0.84, 95% CI 2-sided [0.75 to 0.93]

4. Secondary Outcome: Major Coronary Events Among All Patients Ever Randomized to Simvastatin Plus Ezetimibe Versus All Patients Allocated to Placebo
Description: Major coronary events defined as coronary death or non-fatal myocardial infarction. Myocardial infarction adjudicated based on the presence of serial changes in cardiac biomarkers (e.g. troponin, creatine kinase), typical ECG changes and typical cardiac symptoms. If myocardial infarction was fatal and post-mortem examination findings were available, this information was also assessed. All potential coronary events were adjudicated, using pre-specified objective criteria, by clinicians blinded to study treatment allocation and lipid levels. Numbers provided = number of patients with events.
Time Frame: Median follow-up 4.9 years
Measure: Number; unit: participants
Arm/Group | Simvastatin Plus Ezetimibe | Placebo
Number analyzed (Participants) | 4650 | 4620
participants | 213 | 230
Statistical Analysis 1: Comparison: Simvastatin Plus Ezetimibe vs Placebo; All analyses by intention to treat; Test type: Superiority or Other; p = 0.37, Log Rank; Risk Ratio (RR) = 0.92, 95% CI 2-sided [0.76 to 1.11]

5. Secondary Outcome: Non-hemorrhagic Stroke Among All of Patients Ever Randomized to Simvastatin Plus Ezetimibe Versus All Patients Allocated to Placebo
Description: Stroke was defined as rapid onset of focal or global neurological deficit, with duration greater than 24 hours. Clinical notes and brain imaging were sought to determine the stroke etiology, and if the stroke was fatal and post-mortem examination findings were available, this information was also assessed. All potential stroke events (including transient ischemic attack and intracerebral hemorrhage) were adjudicated, using pre-specified objective criteria, by clinicians blinded to study treatment allocation and lipid levels. Numbers provided = number of patients with events.
Time Frame: Median follow-up 4.9 years
Measure: Number; unit: participants
Arm/Group | Simvastatin Plus Ezetimibe | Placebo
Number analyzed (Participants) | 4650 | 4620
participants | 131 | 174
Statistical Analysis 1: Comparison: Simvastatin Plus Ezetimibe vs Placebo; All analyses by intention to treat; Test type: Superiority or Other; p = 0.01, Log Rank; Risk Ratio (RR) = 0.75, 95% CI 2-sided [0.60 to 0.94]

6. Secondary Outcome: Coronary or Non-coronary Revascularization Among All Patients Ever Randomized to Simvastatin Plus Ezetimibe Versus All Patients Allocated to Placebo
Description: Revascularization included any arterial revascularization procedure, whether surgical or percutaneous, but excluded revascularization performed for hemodialysis vascular access (e.g. fistuloplasty) or to the donor kidney transplant artery. Revascularization included amputations for vascular disease (rather than for trauma or infection). All potential revascularization events (including angiography) were adjudicated, using pre-specified objective criteria, by clinicians blinded to study treatment allocation and lipid levels. Numbers provided = number of patients with events.
Time Frame: Median follow-up 4.9 years
Measure: Number; unit: participants
Arm/Group | Simvastatin Plus Ezetimibe | Placebo
Number analyzed (Participants) | 4650 | 4620
participants | 284 | 352
Statistical Analysis 1: Comparison: Simvastatin Plus Ezetimibe vs Placebo; All analyses by intention to treat; Test type: Superiority or Other; p = 0.0036, Log Rank; Risk Ratio (RR) = 0.79, 95% CI 2-sided [0.68 to 0.93]

7. Secondary Outcome: End-stage Renal Disease Among All Patients Not on Dialysis at the Time of Randomization to Simvastatin Plus Ezetimibe Versus Placebo
Description: End-stage renal disease was defined as initiation of maintenance dialysis or renal transplantation. Temporary dialysis was excluded. All potential dialysis and transplant events were adjudicated, using pre-specified objective criteria, by clinicians blinded to study treatment allocation and lipid levels. Numbers provided = number of patients with events.
Time Frame: Median follow-up 4.9 years
Measure: Number; unit: participants
Arm/Group | Simvastatin Plus Ezetimibe | Placebo
Number analyzed (Participants) | 3117 | 3130
participants | 1057 | 1084
Statistical Analysis 1: Comparison: Simvastatin Plus Ezetimibe vs Placebo; All analyses by intention to treat; Test type: Superiority or Other; p = 0.41, Log Rank; Risk Ratio (RR) = 0.97, 95% CI 2-sided [0.89 to 1.05]

ADVERSE EVENTS:
Time Frame: Median follow-up 4.9 years
Arm/Group | Simvastatin Plus Ezetimibe | Placebo
Serious Adverse Events (participants affected / at risk) | 1142/4650 | 1115/4620
Other Adverse Events (participants affected / at risk) | 992/4650 | 960/4620
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Simvastatin Plus Ezetimibe (N=4650) | Placebo (N=4620)
Vascular death (Vascular disorders) | 361 | 388 — Note that the sum total of vascular deaths, non-vascular deaths and unknown causes of death equates to all cause mortality
Non-vascular deaths (General disorders) | 668 | 612 — Note that the sum total of vascular deaths, non-vascular deaths and unknown causes of death equates to all cause mortality
Unknown causes of death (General disorders) | 113 | 115 — Note that the sum total of vascular deaths, non-vascular deaths and unknown causes of death equates to all cause mortality
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Simvastatin Plus Ezetimibe (N=4650) | Placebo (N=4620)
Muscle pain (Musculoskeletal and connective tissue disorders) | 992 | 960

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes